CLINICAL TRIAL: NCT05085106
Title: A Phase I Study to the Safety, Tolerability, and Pharmacokinetic Characteristics of Felbinac Trometamol Eye Drops of Single-dose and Multiple-dose in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of Felbinac Trometamol Eye Drops
Acronym: Binaprofen
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GZDGZY-BpED-201901
Record Dates: First submitted 2020-10-08; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Eye drop; Safety; Tolerability

STUDY DESIGN:
Intervention Model Description: The study is designed as single dose escalation in the healthy subjects，the subjects are divided from low dose to high dose into 5 single-dose groups of 0.025%, 0.05%, 0.1%, 0.2% and 0.3%, with both male and female subjects in each group.
  The study is designed as multiple dose escalation in the healthy subjects，the subjects are divided into low dose and high dose groups of 0.1% and 0.2% with both male and female subjects in each group.
  The study was designed as double-blind, all the single-dose groups containing 10 subjects except the single-dose group of 0.025% containing 8 subjects，and with 2 placebo controls in each group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Group Ⅰ, give the felbinac trometamol eye drops, 0.025%，1 drop，once. Group Ⅱ, give the felbinac trometamol eye drops, 0.05%，1 drop，once. Group Ⅲ, give the felbinac trometamol eye drops, 0.1%，1 drop，once. Group Ⅳ, give the felbinac trometamol eye drops, 0.2%，1 drop，once. Group Ⅴ, give the felbinac trometamol eye drops, 0.3%，1 drop，once. Multiple Group I, give the felbinac trometamol eye drops, 0.1%，1 drop per time，four times each day, for seven days totally.
  Multiple Group II, give the felbinac trometamol eye drops, 0.2%，1 drop per time，four times each day, for seven days totally.
  Interventions: Drug: Felbinac trometamol eye drop
- Placebo group (Placebo Comparator): Group Ⅰ, give the placebo eye drops, 0.0%，1 drop，once. Group Ⅱ, give the placebo eye drops, 0.0%，1 drop，once. Group Ⅲ, give the placebo eye drops, 0.0%，1 drop，once. Group Ⅳ, give the placebo eye drops, 0.0%，1 drop，once. Group Ⅴ, give the placebo eye drops, 0.0%，1 drop，once. Multiple Group I, give the placebo eye drops, 0.0%, 1 drop per time, four times each day, for seven days totally.
  Multiple Group II, give the placebo eye drops, 0.0%, 1 drop per time, four times each day, for seven days totally.
  Interventions: Drug: Placebo eye drop

INTERVENTIONS:
Drug: Felbinac trometamol eye drop — Felbinac trometamol eye drop: 0.025%、0.05%、0.1%、0.2%、0.3%, 1 drop will be instilled as instructed over one day in single-dose study; 0.1%, 0.2%, 1 drop per time, four times each day and for seven days totally in multiple-dose study.
  Arms: Test group
Drug: Placebo eye drop — Placebo eye drop: 0.0%, 1 drop will be instilled as instructed over one day in single-dose study; 0.0%, 1 drop per time, four times each day and for seven days totally in multiple-dose study.
  Arms: Placebo group

SUMMARY:
To evaluate the safety and tolerability of felbinac trometamol eye drops of single-dose, multiple-dose, dose escalation in healthy subjects, for providing the basis for the dose setting in the later clinical study.

DETAILED DESCRIPTION:
In the single-center, randomized, double-blind, placebo-controlled, single-dose dose escalation study, 48 healthy volunteers will be divided from low dose to high dose into 5 single-dose groups of 0.025%, 0.05%, 0.1%, 0.2% and 0.3%, with both male and female subjects in each group. The study was designed as double-blind, all the single-dose groups containing 10 subjects except the single-dose group of 0.025% containing 8 subjects，and with 2 placebo controls in each group.

Pharmacokinetics blood sampling in different dose groups was designed from low dose to high dose into 4 single-dose groups of 0.05%, 0.1%, 0.2% and 0.3%.

In the single-center, randomized, double-blind, placebo-controlled, multiple-dose dose escalation study, 20 healthy volunteers will be divided into low dose and high dose groups of 0.1% and 0.2%, with both male and female subjects in each group. The study was designed as double-blind, all the dose groups containing 8 subjects and 2 placebo controls.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years old, male or female;
* Weight: Male subjects should not be less than 50.0kg and female subjects should not be less than 45.0kg, BMI within the range of 19.0 and 26.0 kg/m2(Including the threshold);
* Eyes corrected visual acuity should be ≥ 1.0 in both eyes and intraocular pressure, slit lamp and fundus examination were normal or abnormality with no clinical significance;
* The female subjects should be guaranteed to take effective contraception before selected in within a month prior，and all the subjects Regardless of the gender are willing to take effective contraception and no pregnancy is planned for the next 6 months;
* Volunteer to participate in the study and sign informed consent.

Exclusion Criteria:

* With ocular diseases, including a history of inner eye surgery or laser surgery;
* Subjects who had worn contact lenses within 2 weeks prior screening or need to wear it during the study;
* Subjects who had taken any medicine including Eye ophthalmic drug within 2 weeks prior screening；
* Subjects with a history of central nervous, mental, cardiovascular, renal, liver, respiratory, metabolic and musculoskeletal systems;
* Subjects'pretest physical examination, vital signs, ELECTRO cardiogram, laboratory examination and investigator's determination of abnormality with clinical significance.
* The results of eight immunological tests(HBsAg、HBsAb、HBEAG、HABEAB、HbcAb、HCVAb、TPPA、HIV-P24 Antigen/antibody) is abnormality with clinical significance.
* A history of clinically significant allergy, especially drug allergy, allergy to aspirin or other non-steroidal anti-inflammatory drugs or known allergy to the drug component or biphenylacetic acid;
* The average daily smoking amount in the first 3 months was more than 5 cigarettes;
* Alcohol dependence is suspected or confirmed, with alcohol intake averaging more than 2 units per day for 3 months (1 unit =10 mL ethanol, i.e. 1 unit =200 mL beer at 5% alcohol or 25 mL spirits at 40% alcohol or 83 mL wines at 12% alcohol) or alcohol tests positive;
* A history of drug abuse, or positive urine tests for ketamine, morphine, methylamphetamine, dimethylene dioxymethamphetamine, or tetrahydrocannabinic acid;
* Participation in other the clinical trial within 3 months before;
* Blood donation or blood loss ≥400 mL within 3 months before;
* Pregnant or lactating women and those planning to become pregnant;
* Subjects with a history of needle and blood dizziness or intolerance to venipuncture;
* The investigator thinks it is not suitable to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Ophthalmic examination results in single-dose study | 0 hours before administration (within 60 minutes before administration), and 1 hour±10 minutes after administration
  The change of ocular symptoms and signs: baseline (within 60 minutes before administration) and 1 hours±10 minutes after administration
Ophthalmic examination results in multiple-dose study | 0 hours before administration (within 60 minutes before first administration in each day), and 1 hour±10 minutes after each administration
  The change of ocular symptoms and signs: baseline (within 60 minutes before the first dose in each day) and 1 hours±10 minutes after each administration
Ophthalmic examination results in single-dose study | screening period (from Day-14 to Day-1) , 24 hours after administration
  The change of Fundus examination and slit lamp examination: screening period (from Day-14 to Day-1), 24 hours after administration
Ophthalmic examination results in multiple-dose study | screening period (from Day-14 to Day-1) , 48 hours after the last administration
  The change of Fundus examination and slit lamp examination: screening period (from Day-14 to Day-1), 48 hours after the last administration
Ophthalmic examination results in single-dose study | screening period(from Day-14 to Day-1) , 4 hours ± 20minutes after administration
  The change of Fluorescence staining on cornea: screening period (from Day-14 to Day-1), 4 hours ±20 minutes after administration
Ophthalmic examination results in multiple-dose study | screening period(from Day-14 to Day-1) , 4 hours ± 20minutes after the last administration
  The change of Fluorescence staining on cornea: screening period (from Day-14 to Day-1), 4 hours ±20 minutes after the last administration
Intraocular pressure values in single-dose study | screening period(from Day-14 to Day-1) , 24 hours after administration
  The change of Intraocular pressure: Screening period (from Day-14 to Day-1), 24 hours after administration
Intraocular pressure values in multiple-dose study | screening period(from Day-14 to Day-1) , 48 hours after the last administration
  The change of Intraocular pressure: Screening period (from Day-14 to Day-1), 48 hours after the last administration
Visual acuity values in single-dose study | screening period(from Day-14 to Day-1) , 24 hours after administration
  The change of visual acuity: Screening period (from Day-14 to Day-1), 24 hours after administration
Visual acuity values in multiple-dose study | screening period(from Day-14 to Day-1) , 48 hours after the last administration
  The change of visual acuity: Screening period (from Day-14 to Day-1), 48 hours after the last administration
Adverse events (AEs) in single-dose study | All adverse events are collected from the signing of written informed consent up to 24 hours after drug administration.
  The incidence of adverse reactions
Adverse events (AEs) in multiple-dose study | All adverse events are collected from the signing of written informed consent up to 72 hours after the last drug administration.
  The incidence of adverse reactions
Serious adverse events (SAEs) in single-dose study | All serious adverse events are collected from the signing of written informed consent up to 24 hours after drug administration.
  All serious adverse events that occur during the clinical study
Serious adverse events (SAEs) in multiple-dose study | All serious adverse events are collected from the signing of written informed consent up to 72 hours after the last drug administration.
  All serious adverse events that occur during the clinical study

SECONDARY OUTCOMES:
AUC0-t in single-dose study | 0 hour before administration (within 60 minutes before administration) and"10 minutes"，"20 minutes","30 minutes","45 minutes","1 hour ","1.5 hours","2 hours","3 hours","4 hours","6 hours","8 hours","12 hours"and "24 hours"after administration
  the active metabolite biphenylacetic acid in plasma is determined and the pharmacokinetic parameter is calculated.
AUCss0-t in multiple-dose study | 0 hour before the last administration (within 15 minutes) and"10 minutes"，"20 minutes","30 minutes","45 minutes","1 hour ","1.5 hours","2 hours","3 hours","4 hours","6 hours","8 hours","12 hours"and "24 hours"after the last dose (steady state)
  the active metabolite biphenylacetic acid in plasma is determined and the pharmacokinetic parameter is calculated.
Cmax in single-dose study | 0 hour before administration (within 60 minutes before administration) and"10 minutes"，"20 minutes","30 minutes","45 minutes","1 hour ","1.5 hours","2 hours","3 hours","4 hours","6 hours","8 hours","12 hours"and "24 hours"after administration
  the active metabolite biphenylacetic acid in plasma is determined and the pharmacokinetic parameter is calculated.
Cmax in multiple-dose study | 0 hour before the last administration (within 15 minutes) and"10 minutes"，"20 minutes","30 minutes","45 minutes","1 hour ","1.5 hours","2 hours","3 hours","4 hours","6 hours","8 hours","12 hours"and "24 hours"after the last dose (steady state)
  the active metabolite biphenylacetic acid in plasma is determined and the pharmacokinetic parameter is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zhao, Ph.D., Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China